CLINICAL TRIAL: NCT00233571
Title: A Multi-Centre Open Label Continuation Study With Subcutaneous D2E7 (Adalimumab) for Patients With Rheumatoid Arthritis Who Completed a Preceding Clinical Study With D2E7 (Adalimumab)
Brief Title: A Long Term Roll-over Study to Investigate the Efficacy and Safety of Adalimumab Given Long-term to Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DE018
Record Dates: First submitted 2005-09-13; First posted 2005-10-06 (Estimated); Last update posted 2011-11-22 (Estimated); Status verified 2011-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab; Injections, Subcutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adalimumab 40mg subcutaneous (SC) every other week (EOW) (Experimental): Adalimumab 40mg subcutaneous (SC) every other week (EOW)
  Interventions: Biological: Adalimumab 40 mg subcutaneous (SC) every other week (EOW)

INTERVENTIONS:
Biological: Adalimumab 40 mg subcutaneous (SC) every other week (EOW)
  Other Names: ABT-D2E7; adalimumab; Humira

SUMMARY:
The purpose of the study is to assess the long-term safety and clinical efficacy of adalimumab in patients with rheumatoid arthritis

ELIGIBILITY:
Inclusion Criteria:

* Completion of a previous D2E7 study
* Subject is in good health (Investigator discretion) with a recent stable medical history

Exclusion Criteria:

* Former enrollment in this trial (DE018)
* Subject is considered by the investigator, for any reason, to be an unsuitable candidate for the study
* Female subject who is pregnant or breast feeding or considering becoming pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 796 (Actual)
Dates: Start 2000-06; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Clinical response indicators | 5 years

SECONDARY OUTCOMES:
Safety parameters | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Hartmut Kupper, MD, Study Director — Abbott